CLINICAL TRIAL: NCT07108478
Title: A Prospective, Multicenter, Observational Study of the Safety and Efficacy of Emergency Transcatheter Aortic Valve Replacement in Patients With Severe Aortic Stenosis
Acronym: E-TAVR-2025
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Chuanbao Li, Clinical Professor, Qilu Hospital of Shandong University
Other Study IDs: KYLL-202503-007-1
Record Dates: First submitted 2025-07-01; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: Severe Aortic Valve Stenosis; TAVR; emergency
MeSH Terms: conditions — Aortic Valve Stenosis; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case
  Interventions: Device: Transcatheter aortic valve and recyclable delivery system

INTERVENTIONS:
Device: Transcatheter aortic valve and recyclable delivery system — In this study, the transcatheter aortic valve and its recycling delivery system were VitaFlow Liberty®, a TAVR product independently developed by Shanghai Minimally Invasive Cardiovascular Treatment Co., Ltd. (approved and marketed by NMPA). This product is equipment/consumables routinely purchased by hospitals. For routine clinical use, it is designed for transcatheter aortic valve implantation. The valve is delivered to the intended implantation site via the peripheral artery by retrograde flow through the delivery system, realizing the delivery, positioning and release of the valve. Under the supervision of medical imaging equipment, the valve is delivered to the lesion site of the aortic valve, and marked by the diseased aortic annulus, to release the valve and relieve the stenosis at the lesion site, thereby ensuring smooth aortic flow, improving cardiac function and achieving therapeutic purposes.

SUMMARY:
The research name of this project is: A prospective, multicenter and observational study on the safety and effectiveness of emergency transcatheter aortic valve replacement (TAVR) in the treatment of patients with severe aortic stenosis. It is a prospective, multi-center clinical study, and 35 cases are planned to be enrolled and followed up for 12 months (before discharge, 30 days, 6 months and 12 months). The research instruments used are VitaFlow Liberty® transcatheter aortic valve and recoverable delivery system. The purpose of this study is to evaluate the safety and effectiveness of emergency TAVR in patients with severe aortic stenosis. The main end point is the cumulative all-cause mortality 12 months after operation, and the secondary end points mainly include adverse cerebrovascular events (MACCE), acute renal injury, implantation rate of permanent pacemaker and valve function.

DETAILED DESCRIPTION:
The research name of this project is: A prospective, multicenter and observational study on the safety and effectiveness of emergency transcatheter aortic valve replacement (TAVR) in the treatment of patients with severe aortic stenosis. The prognosis of patients with severe aortic stenosis (AS) is extremely poor in emergency, and the mortality of traditional balloon angioplasty (PBAV) is high. As a new treatment method, emergency TAVR needs multi-center data to verify its safety and effectiveness. Based on the preliminary results of a single center, this study was extended to multiple centers in China, aiming at providing high-level evidence, helping to optimize the implementation strategy of emergency TAVR, and promoting its wide application in patients with severe aortic stenosis, thus improving the clinical prognosis and quality of life of patients. This study is a prospective, multi-center clinical study, and 35 patients are planned to be enrolled. All participants are followed up before discharge, 30 days, 6 months and 12 months after valve implantation, and the research unit independently manages data, including data collection, collation and statistical analysis. The research instruments used are VitaFlow Liberty® transcatheter aortic valve and recoverable delivery system. The purpose of this study is to evaluate the safety and effectiveness of emergency TAVR in patients with severe aortic stenosis. The main end point is the cumulative all-cause mortality 12 months after operation, and the secondary end points mainly include adverse cerebrovascular events (MACCE), acute renal injury, implantation rate of permanent pacemaker and valve function. The selection criteria are: patients with severe aortic stenosis diagnosed by medical treatment; Meet one of the emergency TAVR indications (shock, persistent ventricular tachycardia or ventricular fibrillation, unstable angina pectoris or chronic heart failure requiring mechanical circulatory assistance devices, etc.); Voluntary participation and signing of informed consent. The main exclusion criteria are: aortic root anatomy and lesions are not suitable for artificial valve implantation; Anatomical morphology or vascular diseases that affect the instrument approach; Left ventricular outflow tract obstruction; Primary dilated cardiomyopathy; Thrombosis in left ventricle; Patients who cannot receive anticoagulant or antiplatelet therapy, etc. The statistical methods used are descriptive analysis, Kaplan-Meier survival analysis and Cox proportional hazard model (SAS 9.4). Following the Helsinki Declaration, China's Quality Management Standard for Clinical Trials of Medical Devices and ISO 14155:2011, all patients signed informed consent forms with the approval of the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe aortic stenosis diagnosed at the clinic: peak transvalvular flow velocity ≥4.0m/s, or mean transvalvular pressure difference ≥40mmHg(1 mmHg=0.133kPa), or aortic valve orifice area < <0.8cm2 (or effective aortic valve orifice area index < 0.5 cm2/m2);
2. Meet one of the following emergent TAVR indications:

1) Shock; 2) Combined with persistent ventricular tachycardia or ventricular fibrillation; 3) Difficulty in improving unstable angina pectoris or chronic heart failure requiring mechanical circulatory assistance with drugs; 4) Cardiopulmonary resuscitation is required for cardiac arrest; 3. Patients who can understand the purpose of the study, voluntarily participate in and sign the informed consent form, and are willing to accept the relevant examinations and clinical follow-up.

Exclusion Criteria:

1. Aortic root anatomy and lesions are not suitable for prosthetic valve implantation;
2. Anatomic morphology or vascular diseases affecting the instrument approach;
3. Left ventricular outflow tract obstruction;
4. Primary dilated cardiomyopathy;
5. Thrombus in the left ventricle;
6. Patients who are unable to receive anticoagulation or antiplatelet therapy;
7. Allergy to or resistance to Nitinol;
8. Active stage of infective endocarditis or other infection that the researcher believes affects the operation;
9. Severe disability senile dementia;
10. Patients with a life expectancy of less than half a year;
11. The investigator determined that the patient or family had poor compliance or declined to complete the study as required.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 1. Severe aortic stenosis 2, high risk of surgery, or surgical taboo, is not suitable for conventional surgery valve replacement; 3, anatomically suitable for TAVI/TAVR
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative all-cause mortality at 12 months postoperatively | 12 months
  All-cause death includes cardiac death and non-cardiac death

SECONDARY OUTCOMES:
Incidence of major adverse cardiovascular events | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  Incidence of major adverse cardiovascular events (MACCE including mortality, disabling stroke, myocardial infarction, reoperation) calculated as number of occurrences/total number of occurrences
Incidence of acute kidney injury | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  Incidence of acute kidney injury (AKIN Grade 2 or 3, or renal replacement therapy (RRT: hemodialysis, intraperitoneal dialysis, hemofiltration)) calculated as: Occurred/Total
Incidence of permanent pacemaker implantation | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  Incidence of permanent pacemaker implantation, calculated as: Cases Occurred/Total Cases
Incidence of severe vascular complications | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  Incidence of severe vascular complications, calculated as: number of cases/total number of cases
The incidence of other TAVR-related complications | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  The incidence of other TAVR-related complications, including conversion to surgical thoracotomy, accidental cardiopulmonary mechanical assistance, coronary occlusion, ventricular septal perforation, mitral valve damage or loss of function, cardiac tamponade, endocarditis, valve thrombosis, valvular ectopic (shift, embolism, false release), valvular implant, reoperation due to valve dysfunction (TAVR, SAVR, BAV), was calculated as: Cases Occurred/Total Cases
Valve function (assessed by echocardiography) | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  Valve function (assessed by echocardiography): valve function (e.g., aortic valve orifice area, mean pressure differential across the aortic valve), valve regurgitation, perivalvular leakage, moderate or severe valve stenosis
Change in cardiac function (NYHA) | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  NYHA classification: Divided into four levels, Grade I: No discomfort in daily activities, and no restriction in physical activities. Grade II: Mild activity restriction, no symptoms at rest, but daily activities (such as climbing stairs) can cause fatigue and palpitation. Grade III: obvious activity limitation, no symptoms at rest, but slight activity (such as walking) will cause symptoms. Grade Ⅳ: There are symptoms at rest, and any activity aggravates discomfort.
Change in cardiac function (NT-proBNP) | Perioperative/Periprocedural, 30 days, 6 months, 12 months
  NT-proBNP: Secreted by ventricular myocytes when the pressure load of the heart increases (such as heart failure and myocardial stretching), it is the precursor of BNP, obtained by laboratory examination
Success rate of devices, calculation method: number of successful devices/total number of cases | Perioperative/Periprocedural
  calculation method: number of successful devices/total number of cases
Implantation of mechanical circulation assistance device (MCS) | Perioperative/Periprocedural
  Implantation of mechanical circulation assistance device (MCS), calculated as: Cases of mechanical circulation assistance device implantation/Total cases

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodali SK, Thourani VH, Kirtane AJ. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2016 Apr 21;374(16):1591. doi: 10.1056/NEJMc1600179. No abstract available. PMID 27096593
- [Background] Pache G, Schoechlin S, Blanke P, Dorfs S, Jander N, Arepalli CD, Gick M, Buettner HJ, Leipsic J, Langer M, Neumann FJ, Ruile P. Early hypo-attenuated leaflet thickening in balloon-expandable transcatheter aortic heart valves. Eur Heart J. 2016 Jul 21;37(28):2263-71. doi: 10.1093/eurheartj/ehv526. Epub 2015 Oct 7. PMID 26446193
- [Background] Frerker C, Schewel J, Schluter M, Schewel D, Ramadan H, Schmidt T, Thielsen T, Kreidel F, Schlingloff F, Bader R, Wohlmuth P, Schafer U, Kuck KH. Emergency transcatheter aortic valve replacement in patients with cardiogenic shock due to acutely decompensated aortic stenosis. EuroIntervention. 2016 Apr 20;11(13):1530-6. doi: 10.4244/EIJY15M03_03. PMID 25751886
- [Background] Huang H, Kovach CP, Bell S, Reisman M, Aldea G, McCabe JM, Dvir D, Don C. Outcomes of Emergency Transcatheter Aortic Valve Replacement. J Interv Cardiol. 2019 Nov 3;2019:7598581. doi: 10.1155/2019/7598581. eCollection 2019. PMID 31777471
- [Background] Bongiovanni D, Kuhl C, Bleiziffer S, Stecher L, Poch F, Greif M, Mehilli J, Massberg S, Frey N, Lange R, Laugwitz KL, Schymik G, Frank D, Kupatt C. Emergency treatment of decompensated aortic stenosis. Heart. 2018 Jan;104(1):23-29. doi: 10.1136/heartjnl-2016-311037. Epub 2017 May 31. PMID 28566471
- [Background] Block PC, Palacios IF. Clinical and hemodynamic follow-up after percutaneous aortic valvuloplasty in the elderly. Am J Cardiol. 1988 Oct 1;62(10 Pt 1):760-3. doi: 10.1016/0002-9149(88)91218-0. PMID 3421177
- [Background] Buchwald AB, Meyer T, Scholz K, Schorn B, Unterberg C. Efficacy of balloon valvuloplasty in patients with critical aortic stenosis and cardiogenic shock--the role of shock duration. Clin Cardiol. 2001 Mar;24(3):214-8. doi: 10.1002/clc.4960240308. PMID 11288967
- [Background] Grube E, Laborde JC, Gerckens U, Felderhoff T, Sauren B, Buellesfeld L, Mueller R, Menichelli M, Schmidt T, Zickmann B, Iversen S, Stone GW. Percutaneous implantation of the CoreValve self-expanding valve prosthesis in high-risk patients with aortic valve disease: the Siegburg first-in-man study. Circulation. 2006 Oct 10;114(15):1616-24. doi: 10.1161/CIRCULATIONAHA.106.639450. Epub 2006 Oct 2. PMID 17015786
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Carabello BA, Paulus WJ. Aortic stenosis. Lancet. 2009 Mar 14;373(9667):956-66. doi: 10.1016/S0140-6736(09)60211-7. Epub 2009 Feb 21. PMID 19232707
- [Background] Supino PG, Borer JS, Preibisz J, Bornstein A. The epidemiology of valvular heart disease: a growing public health problem. Heart Fail Clin. 2006 Oct;2(4):379-93. doi: 10.1016/j.hfc.2006.09.010. No abstract available. PMID 17448426